CLINICAL TRIAL: NCT02400801
Title: Gonadotropin-releasing Hormone (GnRH) Downregulation Versus Oral Anticonception Prior to ART in Postoperative Endometriosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S55300
Record Dates: First submitted 2015-03-11; First posted 2015-03-27 (Estimated); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Endometriosis; Infertility
Keywords: endometriosis; infertility; assisted reproductive technology
MeSH Terms: conditions — Endometriosis; Infertility | interventions — Triptorelin Pamoate; Ethinyl Estradiol; dienogest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- oral oestroprogestogen pre-treatment (Active Comparator): preparation with oral oestroprogestogens prior to downregulation in an assisted reproductive technology treatment (ART) cycle
  Interventions: Drug: ethinylestradiol + dienogest
- gonadotropin-releasing hormone (GnRH) pre-treatment (Experimental): preparation with gonadotropin-releasing hormone (GnRH) analogues prior to downregulation in an assisted reproductive technology treatment (ART) cycle
  Interventions: Drug: triptorelin

INTERVENTIONS:
Drug: triptorelin — gonadotropin-releasing hormone (GnRH) agonist
  Other Names: decapeptyl
  Arms: gonadotropin-releasing hormone (GnRH) pre-treatment
Drug: ethinylestradiol + dienogest — oral oestroprogestogen
  Other Names: Louise
  Arms: oral oestroprogestogen pre-treatment

SUMMARY:
Does prolonged GnRH downregulation prior to ART improve the clinical pregnancy rate in postoperative endometriosis patients? (A single centre randomised controlled trial)

ELIGIBILITY:
Inclusion Criteria:

* histologically proven endometriosis with complete treatment of all endometriosis lesions during laparoscopy
* only first three ART cycles
* normal uterine cavity
* Eligible for ovarian stimulation with long agonist protocol

Exclusion Criteria:

* FSH>20 IU/L
* presence of large intramural fibroids (> 3 cm)
* <4 oocytes obtained in any previous fresh ART cycle
* ART with sperm derived from testicular biopsy
* ART with Preimplantation Genetic Diagnosis/Screening

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 166 (Estimated)
Dates: Start 2013-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-01-26 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate per initiated ART cycle | participants will be followed for the duration of the ART cycle including the pregnancy test, an expected average of 10 weeks in the active comparator group and an expected average of 18 weeks in the experimental group

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M D'Hooghe, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Tomassetti C, Beukeleirs T, Conforti A, Debrock S, Peeraer K, Meuleman C, D'Hooghe T. The ultra-long study: a randomized controlled trial evaluating long-term GnRH downregulation prior to ART in women with endometriosis. Hum Reprod. 2021 Sep 18;36(10):2676-2686. doi: 10.1093/humrep/deab163. PMID 34370858